CLINICAL TRIAL: NCT07001033
Title: Integrative, Resource-oriented Short Term Dance Movement Therapy for Radio-oncological Patients
Brief Title: Dance Movement Therapy for Radio-oncological Patients
Acronym: DANCE-RT-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAU 24-505-B
Record Dates: First submitted 2025-03-03; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Cancer Patients and Physical Activity
Keywords: Dance Movement Therapy (DMT); Breast or Prostate cancer and complementary therapy; immunophenotyping; muscle strength and bioelectrical impedance analysis (BIA); EQ-5D-5L
MeSH Terms: conditions — Motor Activity; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DMT arm (Other): All patients receive a dance movement therapy intervention once a week for 90 minutes over a period of five weeks, which is combined with psychotherapeutic content. The therapy is carried out by one specially trained DMT therapist with experience in radiooncology.
  The structure of the sessions is designed in such a way that there is a 15-minute starting phase with a mindfulness exercise and opening flash, followed by a 50-minute active phase in which special topic are carried out:
  Therapy sessions and topics:
  1. Introduction. Get to know. Encounter.
  2. Body awareness and dealing with one's own limits.
  3. Social relationships. Proud. Becoming aware of your own resources.
  4. "Cage of emotions". Release.
  5. Conclusion. Reflection and transfer to everyday life. Farewell.
  Interventions: Behavioral: Dance Movement Therapy (DMT)

INTERVENTIONS:
Behavioral: Dance Movement Therapy (DMT) — All participants will be invited to five group meetings at weekly intervals. Each of these therapy sessions will take place with a specific theme. In weeks 1 and 5, data important for the study will be collected once before the short-term DMT and once again at the end of the study. This includes different assessments, laboratory blood tests as well as immunophenotyping. Additionally, patients are requested to complete a questionnaire that addresses QoL. Specific examinations, such as testing the maximal handgrip strength, a BIA and recording Eastern Cooperative Oncology Group (ECOG) performance status are implemented in each of the five meetings.

SUMMARY:
Dance-RT-01 investigates the feasibility and effects of Integrative, resource-oriented short term Dance Movement Therapy (DMT) in radio-oncological patients shortly after radiotherapy (RT). The study assesses clinical outcomes, including reduction of fatigue, improvement of quality of life (QoL), functional capacity and body composition. Immunophenotyping and laboratory blood analyses ensure objectively measurable results. Eligible patients participate in short term DMT, that is combined with psychotherapeutic elements. The trial aims to evaluate DMT's potential as a complementary therapy method in cancer care to support recovery and provide a comprehensive understanding of the therapy's effects.

DETAILED DESCRIPTION:
The study is designed as investigator-initiated, prospective, non-randomized feasibility trial and includes radio-oncological patients (ECOG 0-2) who recently completed RT. The primary endpoint is to decide upon the feasibility, as well as identification of specific immunological changes in peripheral blood that contribute to the success of DMT (longitudinal analysis). The benefit for patients is seen in a resource activation after RT and improvement of well-being. Secondary endpoints include functional capacity, measured by maximum grip strength, body composition, assessed through bioelectrical impedance analysis (BIA), assessment of QoL, pain and reduction of fatigue using validated and standardized questionnaires for patient reported outcomes with comparable results. In addition, immunophenotyping is performed. Further laboratory analyses include inflammatory markers, hormone levels, and nutritional biomarkers. These data are analyzed to evaluate correlation of immunological changes with clinical outcomes.

Participants complete five weekly DMT sessions (90 minutes each). Each session integrates structured movement exercises, music, and psychotherapeutic elements, that can be tailored depending on each individual patient. The therapy is carried out by a certified therapeutic dance instructor with expertise in radio-oncology.

ELIGIBILITY:
Inclusion Criteria:

* Male and female oncological patients
* Age at least 18 years. No upper age limit
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Written informed consent for participation in the study
* Prior RT received shortly before study inclusion (therapy completed)
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including

Exclusion Criteria:

* Inability to speak and understand German
* Serious concurrent neurologic or psychiatric disorders: dementia, uncontrolled seizures, psychosis, schizophrenia, neurosis, autism that would interfere with cooperation with the requirements of the trial
* Familial, sociological, or geographical condition that would preclude study compliance (these conditions should be discussed with the patient before registration in the study)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the study team
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-02-22 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Primary objective | in the week 1 (baseline) in the week 3, in the week 5 (end of study)
  Questionnaire-based (EQ-5D-5L) measurement of well-being containts two main parts: 1) descriptive part in 5 dimentions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimensions have 5 possible answers: no problems, slight problems, moderate problems, severe problems, extreme problems. This is used to define so-called EQ-5D Health States. A total of 3125 different health states can be recorded. Depending on the level, each dimension is assigned a number, resulting in a 5-digit number combination.
  This 5-digit number can be converted into a score (EQ-5D-5L Index) using a special algorithm that is not publicly available and represents the patient's state of health. An index value of 1 represents the best possible state of health, whil 2) Visual Analogue Scale (VAS) a vertical scale on which the participants indicate their self-related state of health, with 0 representing "The worst health you can imagine" and 100 "The best health you can imagine".

SECONDARY OUTCOMES:
Assessment of muscle strength using the Jamar hand dynamometer | weekly: in the week 1 (baseline) 2, 3, 4 and 5 (end of study)
  The subject holds the dynamometer in one hand in line with the forearm and hanging by the thigh. Maximum handgrip strength is then determined without swinging the arm. It is necessary to use the dominate hand for this measurement, because this may help for the interpretation of results.
  The best of three trials is recorded. The dynamometer must be adjusted for hand size, how successfully this is done will affect the accuracy of the measurement. The values in the standard table (in kg) give a guide to scores expected for adults. They are the average of the best scores of the hand.
Assessment of Body Mass Index | weekly: in the week 1 (baseline) 2, 3, 4 and 5 (end of study)
  Following parameter will be measured:
  • Body Mass Index [kg/m²] (BMI) including BMI classification
Assessment of percentage proportion in the patient´s body of fat and skeletal muscle using Bioelectrical Impedance Analysis (BIA) | weekly: in the week 1 (baseline) 2, 3, 4 and 5 (end of study)
  A BIA may provide a non-invasive, rapid method for the assessment of body compartments. For the measurement of a subject, the arms of the subject need to be raised horizontally with the elbows extended and the arms straight at a 90° angle to one's body, holding the display unit. All measurements are performed after the subject had been in supine position for several minutes. All values for the ECW, ICW and TBW compartments are obtained by using the instrument's software option for water volume analysis.
  Following parameters will be measured:
  * Body Fat Percentage [%]
  * Skeletal Muscle Percentage [%]
Assessment of Resting Metabolism (RM) using Bioelectrical Impedance Analysis (BIA) | weekly: in the week 1 (baseline) 2, 3, 4 and 5 (end of study)
  A BIA may provide a non-invasive, rapid method for the assessment of body compartments. For the measurement of a subject, the arms of the subject need to be raised horizontally with the elbows extended and the arms straight at a 90° angle to one's body, holding the display unit. All measurements are performed after the subject had been in supine position for several minutes.
  Following parameters will be measured:
  • Resting Metabolism (RM) [kcal]
Assessment of laboratory parameters and comparison with standard values | in the week 1 (baseline) in the week 3, in the week 5 (end of study)
  complete blood count and white blood cell differential: Erythrocytes (x 10^6/µl , normal: 3.9 - 5.2), haematocrit (%, normal: 35 - 46), haemoglobin (g/dl 11.8 - 15.5), RDW (%, 11.6 - 16.2), MCH (pg, 26 - 33), MCHC (g Hb/dl, 32 - 36), MCV (fl, 81 - 98), MPV (fl, 7.8 - 11)
  All x 10^3/µl normal value in ( ) Leukocytes (4 - 11), basophils (0 - 0.1), eosinophils (0 - 0.5), lymphocytes (1 - 3.5), monocytes (0.1 - 0.9), neutrophils (6 - 7.8)
  C-Reactives proteine (mg/l, normal: <5), gamma-GT (U/l, normal: <40), ferritin (ng/ml, normal: 22-300) , cortisol in serum (µg/dl, normal: 5-25), TSH (mlU/l, normal:0.3-4.00) 25-OH-Vitamin D3 (ng/ml, normal: 30.0-70.0), , vitamin B12 (pg/ml, normal: 211-911), folic acid (ng/ml, normal: 3.89 - 20.0)
Immunophenotyping-longitudinal immunological measurements using flow cytometry | in the week 1 (baseline) in the week 3, in the week 5 (end of study)
  main immune cell populations: granulocytes, monocytes, NK cells, dendritic cells, T and B cells (all counts per µl of blood)
Assessment of the side effects of oncological therapy using NCI CTCEA 5.0 | in the week 1 (baseline) in the week 3, in the week 5 (end of study)
  Assessment according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Translational Radiobiology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No